CLINICAL TRIAL: NCT01185197
Title: Myfortic® Combined With Low-dose Steroid in Minimal Change Nephrotic Syndrome
Brief Title: Myfortic® for Minimal Change Nephrotic Syndrome (MCNS): a Randomized Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Novartis-ST-03
Record Dates: First submitted 2010-08-13; First posted 2010-08-19 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Nephrosis, Lipoid
Keywords: Minimal Change Nephrotic Syndrome; Corticosteroid; Mycophenolate; Remission; Safety
MeSH Terms: conditions — Nephrosis, Lipoid | interventions — Mycophenolic Acid; Steroids; Prednisolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Myfortic plus low-dose steroid (Experimental): Not necessary
  Interventions: Drug: Myfortic plus low-dose steroid
- Standard-dose steroid (Active Comparator): Not necessary
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Myfortic plus low-dose steroid — Prednisolone: 0.25 mg/kg/day for 8 weeks then 0.15 mg/kg/day for 8 weeks then 0.1 mg/kg/day for 8 weeks then off Myfortic: 720 mg b.i.d. (540 mg b.i.d. if body weight less than 60 kg) for 24 weeks then off
  Other Names: Mycophenolate sodium
  Arms: Myfortic plus low-dose steroid
Drug: Prednisolone — 1 mg/kg/day to be tapered over a period of 24 weeks at the discretion of the attending physician
  Arms: Standard-dose steroid

SUMMARY:
Study objective: To investigate the potential therapeutic efficacy of enteric-coated mycophenolate sodium combined with low-dose corticosteroid as first-line treatment for minimal change nephrotic syndrome (MCNS).

DETAILED DESCRIPTION:
This is a prospective, open-label, randomized study in which patients who present for the first time with a clinical diagnosis of idiopathic MCNS proven on renal biopsy will be assigned to either conventional standard-dose prednisolone monotherapy or myfortic combined with low-dose prednisolone treatment for 6 months. Clinical response and relapse rates within 6 months of treatment cessation will be the main outcome parameters.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 - 65 years of age
* First histologic diagnosis of MCNS
* Proteinuria > 3.5 g/day
* Patients who are willing to give written, informed consent

Exclusion Criteria:

* Presence of secondary causes of MCNS
* History of glomerular disease including MCNS
* eGFR < 50 ml/min/1.73m2
* Renal histology showing pathologies other than MCNS
* Female of child-bearing age who are unwilling to practice effective contraception
* Patients simultaneously participating in another study or who have participated in another study within the last 30 days of entry into this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Complete remission (24 hour urine protein < 0.3 g) | at 6 months

SECONDARY OUTCOMES:
Occurrence of cushingoid facies, striae, acne, weight gain, GI disturbance, cytopenia, infection | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sydney CW Tang, MD, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China

REFERENCES:
- [Derived] Azukaitis K, Palmer SC, Strippoli GF, Hodson EM. Interventions for minimal change disease in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2022 Mar 1;3(3):CD001537. doi: 10.1002/14651858.CD001537.pub5. PMID 35230699
- [Derived] Ma MKM, Yap DYH, Li CL, Mok MMY, Chan GCW, Kwan LPY, Lai KN, Tang SCW. Low-dose corticosteroid and mycophenolate for primary treatment of minimal change disease. QJM. 2020 Jun 1;113(6):399-403. doi: 10.1093/qjmed/hcz297. PMID 31769845